CLINICAL TRIAL: NCT06980974
Title: Quasi-Randomized Controlled Trial of Acceptance and Commitment Therapy for Chemsex
Brief Title: Acceptance and Commitment Therapy for Chemsex
Acronym: ACT-for-chemse
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not received.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicholas C. Borgogna, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300014764
Record Dates: First submitted 2025-04-21; First posted 2025-05-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chemsex
Keywords: chemsex; ACT
MeSH Terms: conditions — Chemsex | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-for-chemsex (Experimental): 16 weeks of ACT to reduce chemsex
  Interventions: Behavioral: ACT-for-chemsex
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: ACT-for-chemsex — 16 weeks of acceptance and commitment therapy, delivered online weekly, 45-55 minute sessions
  Arms: ACT-for-chemsex
Other: Treatment as Usual (TAU) — Participants in TAU will receive health/mental health interventions as needed
  Arms: Treatment as usual

SUMMARY:
Quasi-randomized control trial of acceptance and commitment therapy (ACT) for chemsex.

DETAILED DESCRIPTION:
Intervention will entail a prescreening, intake session, 16 therapy sessions, and a six-month follow-up. Each session will be 45-55 minutes long. Participants in ACT-for-chemsex will be compared to participants in a treatment as usual condition.

ELIGIBILITY:
Inclusion Criteria:

* Male
* age 18-65
* access to internet capable smart device
* documentation of Alabama residence
* access to a private area to attend tele ACT-for-chemsex sessions
* self-reported chemsex within six-months of intake
* English fluency.

Exclusion Criteria:

* Psychotic disorder
* bipolar disorder
* eating disorder
* major neurocognitive disorder diagnosis
* self-harm or suicide attempt within 12 months of screener
* suicide plan/intention at time of screening
* ongoing treatment for a complex medical comorbidity (e.g., in patient cancer treatment)
* current enrollment in an individual ACT-based psychotherapy intervention.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male (as assigned at birth)
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Chemsex frequency | Baseline, 16 week post-treatment, six month follow-up
  Self-reported chemsex frequency in the past six months

SECONDARY OUTCOMES:
Modified NIDA ASSIST | Baseline, 16 week post-treatment, six month follow-up
  Past six month substance use on the following scale 0=never
  1. Once or Twice
  2. Monthly
  3. Weekly
  4. Daily or Almost Daily
Sexual Health History | Baseline
  Questions will inquire about STI status including a lifetime history and past 12-month diagnostic status for the following STIs: HIV, Gonorrhea, Syphilis, Chlamydia, Hepatitis C, and Genital Herpes. Participants will be asked "In the past year, have you taken PrEP (pre-exposure prophylaxis)?" ("0=No", "1=Yes, Daily PrEP", "2=Yes, On-Demand [2-1-1] PrEP", "3=Yes, Long-acting PrEP", "4=Not sure"). We will include ad-hoc measures commonly used in previous studies for single item assessments of lifetime, past year, past month, and past week number of partnered sexual experiences, sexual partners, and age of first partnered sexual experience. We will also include the ID Risk Behavior (BRAID) scale (e.g., "Had unprotected [no condom] sex with someone who was a one-night stand or someone you had just met?" "yes", "no"), sexual violence questions as recommended by the Centers for Disease Control and Prevention YRCSS standard national questionnaire.
Center for epidemiologic studies depression scale | Baseline, 16 week post-treatment, six month follow-up, every two weeks.
  A series of questions asking about depression symptoms (e.g. " I was bothered by things that usually don't bother me ")
  On the following scale:
  0=Rarely or none of the time (less than 1 day)
  1. Some or a little of the time (1-2 days)
  2. Occasionally or a moderate amount of the time (3-4 days)
  3. Most or all of the time (5-7 days)
generalized anxiety disorder-7 | Baseline, 16 week post-treatment, six month follow-up, every two weeks
  Anxiety measure.
  Over the last two weeks, how often have you been bothered by the following problems?
  e.g. "Feeling nervous, anxious, or on edge"
  0=not at all
  1. several days
  2. more than half the days
  3. nearly every day
Experiential Avoidance Rating Scale | Baseline, 16 week post-treatment, six month follow-up
  A series of questions asking about experiential avoidance symptoms (e.g. "I have gone to extremes to get rid of thoughts I don't like.")
PSY Flex | Through study completion, an average of one a week"
  A series of questions asking about psychological flexibility (e.g. "Even if I am somewhere else with my thoughts, I can focus on what's going on in important moments.")
Patient Checklist-5 | Baseline, 16 week post-treatment, six month follow-up
  A series of questions asking about PTSD symptoms (e.g. " Repeated, disturbing, and unwanted memories of the stressful experience? ")
Quality of Life Scale | Baseline, 16 week post-treatment, six month follow-up
  A series of questions asking about quality of life (e.g. " Relations with parents, siblings, other relatives")
Multidimensional Psychological Flexibility Inventory | Baseline, 16 week post-treatment, six month follow-up
  A series of questions asking about psychological flexibility (e.g. " I was receptive to observing unpleasant thoughts and feelings without interfering with them.")

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with the research community for secondary analysis. Data can be accessed by emailing the PI.
Supporting Information: Analytic Code
Time Frame: 1/1/2031 - 1/1/2035
Access Criteria: Researchers affiliated with Academic institutions.